CLINICAL TRIAL: NCT00943579
Title: Kuvan® (Sapropterin) as a Treatment for Autistic Disorder: An Open Label Extension Protocol
Brief Title: Open-Label Extension Study of Kuvan for Autism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Children's Health Council (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Glen R. Elliott, Chief Psychiatrist and Medical Director, The Children's Health Council
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHC-0902
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Autistic Disorder
Keywords: autism; autistic disorder; tetrahydrobiopterin; sapropterin; treatment
MeSH Terms: conditions — Autistic Disorder | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kuvan® (Experimental): Kuvan® (sapropterin) will be administered to all subjects at 20 mg/kg/day for 16 weeks.
  Interventions: Drug: Kuvan®

INTERVENTIONS:
Drug: Kuvan® — Brand-name Kuvan® (sapropterin) will be administered to all subjects at a dose of 20 mg/kg/day for 16 weeks.
  Other Names: sapropterin; tetrahydrobiopterin

SUMMARY:
This is an open-label extension study available only to subjects who completed an earlier double-blind, placebo-controlled study of sapropterin in children with autism.

DETAILED DESCRIPTION:
This is an open-label extension study available only to subjects who completed an earlier double-blind, placebo-controlled study of sapropterin in children with autism. During this protocol, all subjects will be receiving brand-name Kuvan 20 mg/kg/day for 16 weeks; subject who complete the first 16 weeks will have the option of continuing on Kuvan at the same dose for up to 90 days after the last subject has completed the first 16 weeks of this protocol. The purpose of the study primarily is to gather additional information on safety and efficacy in this population.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have completed earlier trial, CHC 0901 (NCT00850070)
* Parents must be willing and able to sign informed consent

Exclusion Criteria:

* Child failed to complete CHC 0901 (NCT00850070)

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen R Elliott, PhD, MD, Principal Investigator — The Children's Health Council
Locations (1):
- The Children's Health Council, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment spanned from 08/09 - 10/11. Only individuals who completed 0901 (NCT00850070) were eligible to participate in this study thus recruitment was restricted to those already enrolled in that trial. When participants were at their 12-week visit for 0901 (NCT00850070) they were asked if they wanted to continue in the open label extension.
Pre-assignment Details: All participants who consented went straight from the randomized control trial in 0901 (NCT00850070) to entering this trial. No washout period was needed. No participants were excluded who had completed the previous trial.
Groups:
- Kuvan Following Placebo: Kuvan® (sapropterin) will be administered to all subjects at 20 mg/kg/day for 16 weeks. Participants in this arm received Kuvan following the randomized control trial in which they were on placebo.
- Kuvan Following Active Treatment: Kuvan® (sapropterin) will be administered to all subjects at 20 mg/kg/day for 16 weeks. Participants in this arm received Kuvan following the randomized control trial in which they were on active medication.
Period: Overall Study
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Started | 21 | 20
Completed | 15 | 15
Not Completed | 6 | 5
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 20 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5 (1) | 5 (1) | 5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impressions Scale
Description: This is a summary judgment made by a trained clinician based on observed and reported behaviors of the child compared to baseline. It is a 7-point scale (1) very much improved, (2) much improved, (3) minimally improved (4) no change, (5) minimally worse, (6) much worse and (7) very much worse. Chi-square analyses were used to assess change in CHI-I scores (by group, post-test)Mixed-effects regression models determined the main effects attributed to differences by group (BH4 and placebo), time (treated as categorical at levels baseline, 8 weeks, and 16 weeks) and the group-by-time interaction. The mixed-effects models accounted for each participant's outcome data at each time point. The mixed-effects regression model is robust to data dependency that occurs with the repeated assessments of individuals over time & can handle missing data. We used random intercept and trend modeling that accounts for each individual's initial level of symptom severity/functioning and rate of change/time
Time Frame: 16 weeks
Population: The number of participants analyzed included those who completed the open label extension of this study.
Measure: Number; unit: # participants much - very much improved
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 15 | 15
# participants much - very much improved | 3 | 3
Statistical Analysis 1: Comparison: Kuvan Following Placebo vs Kuvan Following Active Treatment; Chi-square analyses were used to assess CGI-I scores. there were no transformations; Test type: Superiority or Other; p > .05, Chi-squared

2. Secondary Outcome: Vineland Adaptive Behavior Scale, 2nd Edition
Description: The Vineland-2 is semi-structured interview designed to communication, daily living, socialization and motor skills. The Vineland-2 is comprised of a total Adaptive Composite Scale; we chose to use 10 subscales that specifically address functional domains relevant for a young ASD sample - Receptive Communication, Expressive Communication, Personal Daily Living Skills, Domestic Daily Living Skills, Community Daily Living Skills, Interpersonal Relations, Play Skills, Coping Skills, Gross Motor Skills, Fine Motor Skills. The scales generate raw or sum, V-, and age-equivalent scores; raw scores were selected for use in this study. Higher subscale scores indicate more skills. Raw scores can range from 0 to 766 for the overall adaptive behavior composite. Subscales are combined to form the overall Adaptive Behavior Composite, which is essentially a weighted average of the various subscales combined.
Time Frame: Weeks baseline (week 16 from CHC-0901), 8 and 16. Primary outcome assessment looked at change between baseline (week 16 from CHC-0901 and week 16 of CHC-0902).
Population: All participants who completed the open label extension were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 15 | 15
units on a scale | 275 (10.77) | 321 (10.78)

3. Secondary Outcome: Children's Yale Brown Obsessive Compulsive Scale
Description: The C-YBOCS is a scale is designed to rate the severity of obsessive and compulsive symptoms in children and adolescents, ages 6 to 17 years. It can be administered by a clinican or trained interviewer in a semi-structured fashion. In general, the ratings depend on the child's and parent's report; however, the final rating is based on the clinical judgement of the interviewer. Rate the characteristics of each item over the prior week up until, and including, the time of the interview. Scores should reflect the average of each item for the entire week, unless otherwise specified.
Time Frame: Weeks 8 & 16
Population: The data was not analyzed secondary to lack of significant findings in primary outcome measures and limited data collected on this measure. The data cannot now be provided as the research team has since disbanded and it is not possible to reanalyze the data at this time.
Arm/Group | Kuvan®
Number analyzed (Participants) | 0

4. Secondary Outcome: Parental Global Assessment
Description: this is a measure of parents impression of improvement.
Time Frame: Weeks 8 & 16
Population: the data were not analyzed secondary to lack of findings in primary outcome measure as well as the nature of an open label study. The data cannot now be provided as the research team has since disbanded and it is not possible to reanalyze the data at this time.
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Preschool Language Scale, 4th Edition (PLS-4)
Description: Measures expressive & receptive language and total scores in ages 0 to 6 years 11 months. The scales generate raw, standard, and age-equivalent scores; raw scores for the total scale were selected for use in this study. Total is average of subscales. Minimum raw score = 0, maximum = 130. Higher raw scores indicate better language skills. Mixed-effects regression models via SPSS MIXED determined the main effects attributed to differences by group (BH4 and placebo), time (treated as categorical at levels baseline, 8 weeks, and 16 weeks) and the group-by-time interaction. The mixed-effects models accounted for each participant's outcome data at each time point. We used random intercept & trend modeling that accounts for each individual's initial level of symptom severity/functioning & rate of change/time
Time Frame: as for outcome 2
Population: All participants completed the open label extension were analyzed in the study.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 15 | 15
units on a scale | 57.24 (5.48) | 77.83 (5.27)

6. Secondary Outcome: Connor's Preschool ADHD Questionnaire
Description: This is a measure of behavioral symptomatology in children 2-6 years of age. The ADHD scale is one subdomain.
Time Frame: Weeks 8 & 16
Population: Data was not analyzed secondary to lack of significant findings in primary outcome measure and reduced number of completed questionnaires. The data cannot now be provided as the research team has since disbanded and it is not possible to reanalyze the data at this time.
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Aberrant Behavior Checklist (ABC)
Description: This is a 58-item informant-based, factor-analyzed scale comprised of a total scale and 5 subscales that generate raw scores. Scores based on a likert scale ranging from 0-3 where 0 is not a problem to 3 where the problem is severe. Subscales include: Irritability, Social Withdrawal, Stereotypic Behaviors, Hyperactivity and Inappropriate Speech. Total maximum score is 174. Higher subscale scores indicate more symptoms. Scores are totaled to compute subscale scores. Mixed-effects regression models via SPSS MIXED determined the main effects attributed to differences by group (BH4 and placebo), time (treated as categorical at levels baseline, 8 weeks, and 16 weeks) and the group-by-time interaction. The mixed-effects models accounted for each participant's outcome data at each time point. We used random intercept and trend modeling that accounts for each individual's initial level of symptom severity/functioning and rate of change/time
Time Frame: as for outcome 2
Population: all participants who completed the open label extension were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 15 | 15
units on a scale | 16.84 (1.68) | 9.70 (1.73)

8. Secondary Outcome: Adverse Events Reporting
Description: This is not a standardized measure but instead a set of questions, both closed and open ended, asked of families about their child's response to the medication. Used for determining whether treatment needed to be discontinued.
Time Frame: Cummulative throughout study
Population: Data were not specifically analyzed but used instead to determine whether treatment needed to be discontinued. The data cannot now be provided as the research team has since disbanded and it is not possible to reanalyze the data at this time.
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the length of the study, i.e., 16 weeks.
Description: All participants were asked at each visit regarding adverse events. Specific examples were asked, such as difficulties with sleep, irritability and bowel movements then it was left open ended for parents to describe if other adverse events were noted.
Arm/Group | Kuvan Following Placebo | Kuvan Following Active Treatment
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 14/21 | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kuvan Following Placebo (N=21) | Kuvan Following Active Treatment (N=20)
Changes in bowel movements (Gastrointestinal disorders) | 5 | 5 — Diarrhea
Irritability (Psychiatric disorders) | 3 | 4 — Increased irritability in a variety of settings
Difficulty Sleeping (Nervous system disorders) | 6 | 5 — Persistent changes in sleep, including onset insomnia, frequent wakening during the night, lightening of sleep
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 — Viral or autoimmune rash
Hyperactivity (Nervous system disorders) | 3 | 0 — Persistent increase in overall activity level in a variety of settings
Anxiety (Psychiatric disorders) | 2 | 0 — Increase in anxious symptoms
Repetitive Behaviors (Nervous system disorders) | 3 | 5 — Sustained changes in or appearance of stereotypies or other odd, repetitive behaviors

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No